CLINICAL TRIAL: NCT02921048
Title: Effects of Omega-3 Fatty Acids in Ambient Air Pollution Exposure in Healthy Adults
Acronym: PISCES
Status: Completed | Type: Observational
Sponsor: U.S. EPA Human Studies Facility (U.S. Federal Agency)
Responsible Party: Principal Investigator, Haiyan Tong, Research biologist, U.S. EPA Human Studies Facility
Other Study IDs: HSF-001
Record Dates: First submitted 2016-09-28; First posted 2016-09-30 (Estimated); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Health Effects of Ambient Air Pollution
Keywords: Eicosapentaenoic Acid; Docosahexaenoic Acid; Ambient Air Pollution
MeSH Terms: interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- omega-3: individuals voluntarily taking at least 3 g/wk of EPA and DHA from dietary sources including fish oil supplements and ocean fish/shellfish consumption for a period of at least 6 months prior to enrollment in the study
  Interventions: Dietary Supplement: omega-3 fatty acids
- control: individuals who have consumed no more than 1 serving size (4-6 oz)/month of ocean fish/shellfish, or no more than 1 pill/month of fish oil supplement during the 6 month period preceding enrollment

INTERVENTIONS:
Dietary Supplement: omega-3 fatty acids
  Groups: omega-3

SUMMARY:
This observational study recruits healthy individuals who have been routinely taking high amount (at least 3 g/wk) of dietary eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA), and those who don't, and examines the efficacy of dietary EPA and DHA in ameliorating the cardiopulmonary effects of exposure to ambient air pollution.

DETAILED DESCRIPTION:
Purpose: To examine the relationship between blood levels of dietary eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) and cardiopulmonary responses to environmental air pollution in healthy adults. EPA and DHA are two important omega-3 fatty acids that are mainly found in seafoods and fish oils and associated with beneficial effects to human physiology.

Participants: Healthy 35-55 year-old male and female subjects will be screened for their dietary intake of EPA and DHA. Qualified volunteers will be divided into two groups, group 1: individuals voluntarily taking at least 3 g/wk of EPA and DHA from dietary sources including fish oil supplements and ocean fish/shellfish consumption for a period of at least 6 months prior to enrollment in the study; group 2: individuals who have consumed no more than 1 serving size (4-6 oz)/month of ocean fish/shellfish, or no more than 1 pill/month of fish oil supplement during the 6 month period preceding enrollment.

Procedures (Methods): In this observational panel study, subjects will come to the U.S. EPA Human Studies Facility for up to 5 sessions, each consisting of 2 consecutive visit days. The following endpoints will be collected: blood pressure, heart rate variability measurements, blood biomarkers, endothelial cell function, retinal venule and arteriole diameter, and lung function. Air pollution exposure will be assessed using area-specific air quality data derived from local air monitoring stations interfaced with activity monitoring and GPS tracked location for each subject.

ELIGIBILITY:
Inclusion Criteria:

* Aged 25-55 years old healthy male and female (19≤BMI≤30).
* Normal resting ECG. No history of heart arrhythmia.
* Oxygen saturation greater than 96% at the time of physical exam.
* Taking at least 3 grams of EPA and DHA from dietary sources including fish oil supplements and ocean fish/shellfish for a 6 months or longer period of time preceding enrollment in the study; or taking no more than 1 serving size (4-6 oz)/month of ocean fish/shellfish, or no more than 1 pill/month of fish oil supplement during the previous 6 months or longer period of time.

Exclusion Criteria:

* Individuals with a history of acute or chronic cardiovascular disease, such as myocardial infarction.
* Individuals with a history of chronic respiratory disease, such as COPD and asthma.
* Individuals with a history of cancer (possible exception for history of non-melanoma skin cancer).
* Uncontrolled hypertension (≥150 systolic, ≥90 diastolic).
* Individuals who are diabetic (previously diagnosed or with hemoglobin A1c level >6.4%).
* Individuals who are currently smoking (including vaping, or using hookah or e cigarettes) or have a smoking history within 1 year of study (defined as more than 1 pk/yr in the past year) or have a greater than/equal to a 5 pack year smoking history.
* Individuals living with a smoker who smokes inside the house.
* Individuals who are regularly exposed to high levels of vapors, dust, gases, or fumes.
* Individuals who do not understand or speak English.
* Individuals who are taking b-blocker medications.
* Individuals who are taking statins.
* Individuals that are unwilling or unable to maintain their current dietary pattern for the whole study.
* Individuals with bleeding or clotting disorders.
* Individuals who have active allergies.
* Individuals who have an allergy to latex, or skin allergy to tape or electrodes.
* Individuals who are pregnant or attempting to become pregnant.
* Individuals who have unspecified illnesses, which in the judgment of the investigators might increase the risk associated with clinical procedures will be a basis for exclusion.
* Individuals who are currently taking anti-depressants.

Temporary exclusion criteria:

* Individuals who have had recent (within 6 months) abdominal and/or eye surgery, or been diagnosed with any type of hernia, as well as any other contraindications for raised intra-abdominal pressure.
* Individuals who have had an acute respiratory illness within 4 weeks.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy 35-55 year-old male and female subjects
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2016-09-15 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
heart rate variability | Sep. 2016 to Sep 2019

SECONDARY OUTCOMES:
endothelial cell function | Sep. 2016 to Sep 2019
diameters of retinal arteries and veins | Sep. 2016 to Sep 2019
pulmonary function indices | Sep. 2016 to Sep 2019
blood biomarkers | Sep. 2016 to Sep 2019

CONTACTS AND LOCATIONS:
Locations (1):
- EPA Human Studies Facility, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Chen H, Zhang S, Shen W, Salazar C, Schneider A, Wyatt LH, Rappold AG, Diaz-Sanchez D, Devlin RB, Samet JM, Tong H. Omega-3 fatty acids attenuate cardiovascular effects of short-term exposure to ambient air pollution. Part Fibre Toxicol. 2022 Feb 9;19(1):12. doi: 10.1186/s12989-022-00451-4. PMID 35139860
- [Derived] Chen H, Zhang S, Shen W, Salazar C, Schneider A, Wyatt L, Rappold AG, Diaz-Sanchez D, Devlin RB, Samet JM, Tong H. The influence of dietary intake of omega-3 polyunsaturated fatty acids on the association between short-term exposure to ambient nitrogen dioxide and respiratory and cardiovascular outcomes among healthy adults. Environ Health. 2021 Dec 7;20(1):123. doi: 10.1186/s12940-021-00809-9. PMID 34872587
- [Derived] Tong H, Zhang S, Shen W, Chen H, Salazar C, Schneider A, Rappold AG, Diaz-Sanchez D, Devlin RB, Samet JM. Lung Function and Short-Term Ambient Air Pollution Exposure: Differential Impacts of Omega-3 and Omega-6 Fatty Acids. Ann Am Thorac Soc. 2022 Apr;19(4):583-593. doi: 10.1513/AnnalsATS.202107-767OC. PMID 34797737